CLINICAL TRIAL: NCT03639532
Title: Is Ceramic-on-Ceramic THA Superior to Ceramic-on-Highly Cross-Linked Polyethylene THA in Patients Less Than 55 Years Old?
Brief Title: Ceramic-on-Ceramic Versus Ceramic-on-HXLPE THA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ewha Womans University (Other)
Responsible Party: Principal Investigator, Young Hoo Kim, Professor, Ewha Womans University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HXLTHA
Record Dates: First submitted 2018-08-15; First posted 2018-08-21 (Actual); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: Osteoarthritis, Hip; Avascular Necrosis of the Femoral Head; Arthropathy of Hip; Hip Arthr
MeSH Terms: conditions — Osteoarthritis, Hip; Femur Head Necrosis

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- COC (Experimental): for the arthritic hip of the patient, total hip arthroplasty(THA) with ceramic on ceramic(COC) bearing couple is implanted. The group with intervention COC THA.
  Interventions: Procedure: COC THA
- COP (Active Comparator): for the arthritic hip of the patient, total hip arthroplasty(THA) with ceramic on highly cross-linked polyethylene bearing couple is implanted. The group with intervention COP THA.
  Interventions: Procedure: COP THA

INTERVENTIONS:
Procedure: COC THA — standard total hip arthroplasty is done, with ceramic on ceramic for the bearing.
  Arms: COC
Procedure: COP THA — standard total hip arthroplasty is done, with ceramic on highly cross linked polyethylene for the bearing.
  Arms: COP

SUMMARY:
Methods to reduce the revision rate of total hip arthroplasties (THAs) because of wear-related issues are important to examine, particularly because younger patients have a disproportionately high risk of revision. The investigators hoped to follow up patients and see if long-term Harris hip scores and WOMAC scores better in younger patients with a ceramic-on-ceramic (COC) THA compared with those with a ceramic-on-highly-cross-linked polyethylene (COP) THA.

DETAILED DESCRIPTION:
High success rates obtained in the general population have stimulated for total hip arthroplasty (THA) in young and active patients. Although there have been substantial improvements in THA, bearing surface wear and osteolysis are major factors limiting the durability of THAs in young and active patients. During the last decade, alternative bearings have been developed, including highly cross-linked polyethylene (HXLPE) and ceramic-on-ceramic (COC) bearings, with the potential to reduce wear and osteolysis in younger, more active patients.

Despite contemporary cementless THA with COC bearings giving excellent clinical and radiographic outcomes, there is concern about squeaking, fracture of the ceramic head or acetabular insert or fretting and corrosion (trunnionosis). Although HXLPE have been reported to reduce polyethylene wear, there is concerned about a potential decrease in toughness, tensile strength and resistance to the propagation of fatigue cracks in a long-term follow-up.

Several noncomparative studies of COC and COP THA have reported promising results in terms of Harris hip scores, radiographic findings, and survival rates, yet we are aware of no long-term comparative clinical studies with a COC THA and a COP THA in the same younger patients. This study aimed to see if long-term Harris hip scores and Western Ontario and McMaster Universities Osteoarthritis (WOMAC) score better in younger patients with a COC THA compared with those with a COP THA.

ELIGIBILITY:
Inclusion Criteria:

* bilateral end-stage hip arthrosis

Exclusion Criteria:

* inflammatory arthritis, foot and ankle disorders, dementia, stroke history, high dislocation of hip, patients older than 55 years

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 148 (Actual)
Dates: Start 2000-01-01 (Actual); Primary Completion 2003-04-30 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
Harris hip score | 15 years after the intervention
  The Harris Hip Score(HHS) was developed by William H. Harris to assess the results of hip surgery or hip replacement. The standard evaluation applies to various hip disabilities and methods of treatment in adults. The original version of the score was first published in 1969. 100 is the best score, and 0 is the worst possible score. HHS has a subset of pain(44 points), function(47 points), absence of deformity(4 points), and range of motion(5 points)

SECONDARY OUTCOMES:
WOMAC(Western Ontario and McMaster Universities) Scores | 15 years after the intervention
  A tool to evaluate patient function associated with knee. The WOMAC measures five items for pain (score range 0-20), two for stiffness (score range 0-8), and 17 for functional limitation (score range 0-68). The total score is summed from individual sections, and 0 is the best possible score.

REFERENCES:
- [Background] Bansal A, Khatib ON, Zuckerman JD. Revision total joint arthroplasty: the epidemiology of 63,140 cases in New York State. J Arthroplasty. 2014 Jan;29(1):23-7. doi: 10.1016/j.arth.2013.04.006. Epub 2013 May 13. PMID 23680502
- [Background] Kim YH, Park JW, Park JS. The 27 to 29-year outcomes of the PCA total hip arthroplasty in patients younger than 50 years old. J Arthroplasty. 2014 Dec;29(12):2256-61. doi: 10.1016/j.arth.2014.02.011. Epub 2014 Feb 12. PMID 24636903
- [Background] Clohisy JC, Oryhon JM, Seyler TM, Wells CW, Liu SS, Callaghan JJ, Mont MA. Function and fixation of total hip arthroplasty in patients 25 years of age or younger. Clin Orthop Relat Res. 2010 Dec;468(12):3207-13. doi: 10.1007/s11999-010-1468-4. PMID 20668972
- [Background] Adelani MA, Keeney JA, Palisch A, Fowler SA, Clohisy JC. Has total hip arthroplasty in patients 30 years or younger improved? A systematic review. Clin Orthop Relat Res. 2013 Aug;471(8):2595-601. doi: 10.1007/s11999-013-2975-x. Epub 2013 Apr 6. PMID 23564363
- [Background] Kim YH, Park JW, Patel C, Kim DY. Polyethylene wear and osteolysis after cementless total hip arthroplasty with alumina-on-highly cross-linked polyethylene bearings in patients younger than thirty years of age. J Bone Joint Surg Am. 2013 Jun 19;95(12):1088-93. doi: 10.2106/JBJS.L.01211. PMID 23783205
- [Background] Capello WN, D'Antonio JA, Feinberg JR, Manley MT, Naughton M. Ceramic-on-ceramic total hip arthroplasty: update. J Arthroplasty. 2008 Oct;23(7 Suppl):39-43. doi: 10.1016/j.arth.2008.06.003. PMID 18922373
- [Background] Bascarevic Z, Vukasinovic Z, Slavkovic N, Dulic B, Trajkovic G, Bascarevic V, Timotijevic S. Alumina-on-alumina ceramic versus metal-on-highly cross-linked polyethylene bearings in total hip arthroplasty: a comparative study. Int Orthop. 2010 Dec;34(8):1129-35. doi: 10.1007/s00264-009-0899-6. Epub 2009 Nov 1. PMID 19882338